CLINICAL TRIAL: NCT06894602
Title: Association of Ultrasonographic Temporal Artery Lesions and Relapse in Patients With Giant Cell Arteritis
Acronym: ALERT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0371 - ALERT
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Giant Cell Arteritis
Keywords: giant cell arteritis; Ultrasound; follow up; monitoring; OGUS score
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with giant cell arteritis at diagnosis: patients routinely monitored for their disease, and who typically benefit from temporal artery ultrasound as part of their disease. Recruitment will be facilitated by the fact that these are "general population" patients with suspected giant cell arteritis.

SUMMARY:
Ultrasound evaluation of the temporal and axillary arteries is currently well recognized in the field of giant cell arteritis (GCA), a disease primarily affecting medium- and large-caliber vessels. Structural ultrasound abnormalities are now well described in this pathology, but their association with relapse and clinical concordance is unknown. There is currently a follow-up score (the OGUS score) for medium- and large-caliber arteries that could also predict the clinical course of the disease.

DETAILED DESCRIPTION:
Prospective bicentric longitudinal study evaluating the association between ultrasound lesions and clinico-biological relapse in patients with giant cell arteritis.

This is a non-interventional study with patients routinely followed for their pathology and classically benefiting from temporal artery ultrasound as part of their disease. Recruitment will be facilitated by the fact that these will be "general population" patients with suspected giant cell arteritis.

The center will enroll 100 patients. The study will take place over 3 visits, including a clinical, biological and ultrasound examination. Ultrasound will not be blinded to the clinic, so we will only need one examiner in the center.

This is a study in routine care, with no additional costs and no expected constraints. The ultrasound examination will be performed as part of their routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patients meeting ACR 2022 criteria for giant cell arteritis.
* No opposition expressed

Exclusion Criteria:

* Patients unable to understand the protocol, under guardianship or curatorship.
* Patients not affiliated to the French Social Security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with giant cell arteritis at disease diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Relapse according to EULAR 2018 criteria | At 12 months
  Relapse is defined with European League Against Rheumatism recommendations according to major or minor relapse criteria.

SECONDARY OUTCOMES:
Relapse according to EULAR 2018 criteria | At 6 month; at 12 month
  Relapse is defined with European League Against Rheumatism recommendations according to major or minor relapse criteria.
Clinical parameter : Age | At inclusion
  One Clinical parameter is defined with the dichotomised variable : age > 50 years (YES) and age <=50 years (NO)
Other prognostic marker : C-Reactive Protein | At inclusion, At 6 month, At 12 month
  Pronostic markers are defined with C-Reactive Protein (in mg/L)
OMERACT Giant Cells arteritis Ultrasonography Score (OGUS) | At 6 month, at 12 month
  It is a score for ultrasound monitoring of temporal arteries by measuring the intima media complex of 8 vascular sites (common temporal trunk, frontal and parietal branches, axillary arteries). If OGUS score is >= 1, the criteria is YES, if OGUS score < 1, the criteria is NO
C-Reactive Protein | At 6 month, at 12 month
  It is a biological marker expressed in mg/L. If CRP >=10 mg/L, the criteria is YES. If CRF < 10 mg/L, the criteria is NO
Erythrocyte Sedimentation Rate (ESR) | At 6 month, at 12 month
  It is a blood test that can show the inflammation in the body, in mm/hour. If ESR >= 15 mm/h, the criteria is YES. If ESR < 15 mm/h, the criteria is NO.
Clinical parameter : loss of vision | At inclusion
  One Clinical parameter is defined with the sudden loss of vision (YES/NO)
Clinical parameter : claudication of the jaw or tongue | At inclusion
  One Clinical parameter is defined with the claudication of the jaw or tongue (YES/NO)
Clinical parameter : temporal headaches | At inclusion
  One Clinical parameter is defined with the temporal headaches (YES/NO)
Clinical parameter : scalp paresthesia | At inclusion
  One Clinical parameter is defined with the scalp paresthesia (YES/NO)
Clinical parameter : abnormal palpation of the temporal arteries | At inclusion
  One Clinical parameter is defined with the abnormal palpation of the temporal arteries (YES/NO)
Clinical parameter : morning stiffness of shoulders and/or neck | At inclusion
  One Clinical parameter is defined with morning stiffness of shoulders and/or neck (YES/NO)
Biological parameter : temporal artery biopsy | At inclusion
  One biological parameter is defined with positive temporal artery biopsy (YES/NO)
Biological parameter : halo sign on ultrasound | At inclusion
  One biological parameter is defined with halo sign on ultrasound (Present/Absent)
Biological parameter : bilateral axillary involvement | At inclusion
  One biological parameter is defined with bilateral axillary involvement (occlusion or stenosis visualized on ultrasound or CT angio or PET scan or MRI)(Present/Absent)
Biological parameter : aortitis | At inclusion
  One biological parameter is defined with aortitis on PET scans of the thoracic or abdominal descending aorta (Present/Absent)
Biological parameter : Sedimentation rate | At inclusion
  One biological parameter is defined with Sedimentation rate >= 50 mm/hour (YES/NO)
Biological parameter : C-Reactive Protein | At inclusion
  One biological parameter is defined with C-Reactive Protein >= 10 mg/L at the first hour (YES/NO)
Other prognostic marker : hemoglobin | At inclusion, At 6 month, At 12 month
  Pronostic markers are defined with hemoglobin (in g/dL)
Other prognostic marker : leukocytes | At inclusion, At 6 month, At 12 month
  Pronostic markers are defined with leukocytes (in giga/L)
Other prognostic markers : platelets | At inclusion, At 6 month, At 12 month
  Pronostic markers are defined with platelets (in giga/L)
Other prognostic marker : Sedimentation rate | At inclusion, At 6 month, At 12 month
  Pronostic markers are defined with Sedimentation rate (in mm/hour)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Brest, Brest
  - Ch Quimper, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.